CLINICAL TRIAL: NCT02093819
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 416970 in Healthy Male Volunteers in a Partially Randomised, Single-blind, Placebo-controlled Trial, Investigation of Relative Bioavailability of BI 416970 (Open-label, Randomised, Three-way Cross-over) and Assessment of Safety and Exposure of BI 416970 in CYP2C9 Genotyped Volunteers (Open-label, Single-dose)
Brief Title: To Assess Safety, Tolerability and Pharmacokinetics of BI 416970 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1345.1; 2013-003560-31 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-02

CONDITIONS: Healthy

ARMS (1):
- BI 416970 single rising dose part (Experimental): single rising dose given as tablet
  Interventions: Drug: Placebo to BI 416970; Drug: BI 416970

INTERVENTIONS:
Drug: Placebo to BI 416970 — single rising doses
Drug: BI 416970 — single rising doses

SUMMARY:
To investigate the safety and tolerability of BI 416970 and to assess the pharmacokinetics (PK) of single rising doses of BI 416970. A further objective is to assess the influence of CYP2C9 phenotype on the PK of BI 416970.

ELIGIBILITY:
Inclusion criteria:

* Healthy males according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure, Pulse Rate), 12-lead electrocardiogram, and clinical laboratory
* Age 18 to 50 years (incl.)
* Body Mass Index 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Known genotype of CYP2C9 isoenzyme

Exclusion criteria:

* Any finding in the medical examination (including Blood Pressure, Pulse Rate or Electrocardiogram) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside of ranges 90-140 mmHg, diastolic blood pressure outside of ranges 50-90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication
* Diseases of the central nervous system (such as epilepsy), other peripheral neurological disorders or psychiatric disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1345.1.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in eight groups.
Groups:
- Placebo: The medication was administered as a single oral dose (Dose = NA) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 10mg: The medication was administered as a single oral dose (dose = 10 mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 25mg: The medication was administered as a single oral dose (Dose = 25mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 50mg: The medication was administered as a single oral dose (dose = 50mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 100mg: The medication was administered as a single oral dose (Dose = 100mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 200mg: The medication was administered as a single oral dose (Dose = 200mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 400mg: The medication was administered as a single oral dose (Dose = 400mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 600mg: The medication was administered as a single oral dose (Dose = 600mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
Period: Overall Study
Arm/Group | Placebo | BI 416970 10mg | BI 416970 25mg | BI 416970 50mg | BI 416970 100mg | BI 416970 200mg | BI 416970 400mg | BI 416970 600mg
Started | 15 | 6 | 10 | 6 | 6 | 6 | 5 | 6
Completed | 15 | 6 | 10 | 6 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: This subject set included all subjects who were dispensed study medication and were documented to have taken ≥1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 416970 10mg | BI 416970 25mg | BI 416970 50mg | BI 416970 100mg | BI 416970 200mg | BI 416970 400mg | BI 416970 600mg | Total
Number analyzed (Participants) | 15 | 6 | 10 | 6 | 6 | 6 | 5 | 6 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (9.2) | 35.7 (7.9) | 38.9 (8.7) | 34.2 (10.0) | 31.0 (4.6) | 31.2 (12.7) | 34.0 (9.5) | 35.3 (10.9) | 34.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 15 | 6 | 10 | 6 | 6 | 6 | 5 | 6 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events
Description: Percentage of subjects with drug-related adverse events
Time Frame: AEs were recorded throughout the trial
Population: The PKS included 59 subjects of the TS who provided at least 1 value of the endpoints Cmax, AUC0-∞, or AUC0-tz.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BI 416970 10mg | BI 416970 25mg | BI 416970 50mg | BI 416970 100mg | BI 416970 200mg | BI 416970 400mg | BI 416970 600mg
Number analyzed (Participants) | 15 | 6 | 10 | 6 | 6 | 6 | 5 | 6
percentage of participants | 6.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 20.0 | 0.0

2. Secondary Outcome: Cmax (Maximum Measured Concentration of the Analyte in Plasma)
Description: Cmax (maximum measured concentration of the analyte in plasma)
Time Frame: 2 hour (h) before drug administration and 15minutes (min), 30min, 45min, 1h,1h 30min, 1h 45min, 2h, 3h, 4h, 4h 15min, 6h, 7h, 8h, 10h, 12h, 24h, 34h and 48h after drug administration
Population: The PKS included 59 subjects of the TS who provided at least 1 value of the endpoints Cmax, AUC0-∞, or AUC0-tz.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | BI 416970 10mg | BI 416970 25mg | BI 416970 50mg | BI 416970 100mg | BI 416970 200mg | BI 416970 400mg | BI 416970 600mg
Number analyzed (Participants) | 6 | 10 | 6 | 6 | 6 | 5 | 5
nmol/L | 15.2 (66.3) | 44.0 (80.5) | 154 (69.6) | 250 (37.2) | 482 (40.3) | 1060 (70.4) | 1610 (50.2)
Statistical Analysis 1: Comparison: BI 416970 10mg vs BI 416970 25mg vs BI 416970 50mg vs BI 416970 100mg vs BI 416970 200mg vs BI 416970 400mg vs BI 416970 600mg; A power model was used to describe functional relationship between dose and Pk parameters. For the evaluation of dose proportionality,slope parameter (B), a two-sided 90% confidence interval of the slope was calculated. Perfect dose proportionality would correspond to a slope of 1; Test type: Superiority or Other; Slope = 1.1313, 90% CI 2-sided [1.0249 to 1.2376], Standard Error of Mean 0.0633 — Evaluation of dose proportionality - all dose groups. Number of subjects included in the analysis=44
Statistical Analysis 2: Comparison: BI 416970 50mg vs BI 416970 100mg vs BI 416970 200mg vs BI 416970 400mg vs BI 416970 600mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Slope = 0.9568, 90% CI 2-sided [0.7830 to 1.1307], Standard Error of Mean 0.1019 — Evaluation of dose proportionality - dose groups 50mg to 600mg. Number of subjects included in the analysis=28

3. Secondary Outcome: AUC 0-infinity (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: AUC 0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
Time Frame: as for outcome 2
Population: The PKS included 59 subjects of the TS who provided at least 1 value of the endpoints Cmax, AUC0-∞, or AUC0-tz.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 416970 10mg | BI 416970 25mg | BI 416970 50mg | BI 416970 100mg | BI 416970 200mg | BI 416970 400mg | BI 416970 600mg
Number analyzed (Participants) | 6 | 10 | 6 | 6 | 6 | 5 | 5
nmol*h/L | 72.8 (41.5) | 195 (49.8) | 566 (54.0) | 992 (36.1) | 1770 (34.6) | 3970 (61.3) | 6150 (23.2)
Statistical Analysis 1: Comparison: BI 416970 10mg vs BI 416970 25mg vs BI 416970 50mg vs BI 416970 100mg vs BI 416970 200mg vs BI 416970 400mg vs BI 416970 600mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Slope = 1.0732, 90% CI 2-sided [0.9946 to 1.1518], Standard Error of Mean 0.0468 — Evaluation of dose proportionality - all dose groups. Number of subjects included in the analysis=44
Statistical Analysis 2: Comparison: BI 416970 50mg vs BI 416970 100mg vs BI 416970 200mg vs BI 416970 400mg vs BI 416970 600mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Slope = 0.9603, 90% CI 2-sided [0.8174 to 1.1032], Standard Error of Mean 0.0838 — Evaluation of dose proportionality - dose groups 50 mg to 600 mg. Number of subjects included in the analysis 28

ADVERSE EVENTS:
Time Frame: From the first intake of trial medication until the end of trial examination, up to 14 days.
Groups:
- BI 416970 10 mg: The medication was administered as a single oral dose (dose = 10 mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 25 mg: The medication was administered as a single oral dose (dose = 25 mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 50 mg: The medication was administered as a single oral dose (dose = 50 mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 100 mg: The medication was administered as a single oral dose (dose = 100 mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 200 mg: The medication was administered as a single oral dose (dose = 200 mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 400 mg: The medication was administered as a single oral dose (dose = 400 mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- BI 416970 600 mg: The medication was administered as a single oral dose (dose = 600 mg) with a total of about 240 mL water in the standing or sitting position following an overnight fast of at least 10 h.
- Total BI 416970 Treatment: All patients affected by AEs during administration of BI 416970 medication .
- Total Treatment: All patients affected by AEs during entire treatment period.
Arm/Group | Placebo | BI 416970 10 mg | BI 416970 25 mg | BI 416970 50 mg | BI 416970 100 mg | BI 416970 200 mg | BI 416970 400 mg | BI 416970 600 mg | Total BI 416970 Treatment | Total Treatment
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/10 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/45 | 0/60
Other Adverse Events (participants affected / at risk) | 1/15 | 1/6 | 3/10 | 1/6 | 0/6 | 2/6 | 2/5 | 1/6 | 10/45 | 11/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | BI 416970 10 mg (N=6) | BI 416970 25 mg (N=10) | BI 416970 50 mg (N=6) | BI 416970 100 mg (N=6) | BI 416970 200 mg (N=6) | BI 416970 400 mg (N=5) | BI 416970 600 mg (N=6) | Total BI 416970 Treatment (N=45) | Total Treatment (N=60)
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 4 | 4
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes